CLINICAL TRIAL: NCT05098912
Title: The Effectiveness of Polydioxanone Thread Embedding Acupuncture Compared to Manual Acupuncture for Nasolabial Fold Reduction
Brief Title: Comparing Polydioxanone Thread Embedding Acupuncture and Manual Acupuncture for Nasolabial Fold Reduction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Yolanda Teja, Resident Doctor of Medical Acupuncture Study Programme University of Indonesia, Indonesia University, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 21060651
Record Dates: First submitted 2021-10-20; First posted 2021-10-28 (Actual); Last update posted 2022-02-09 (Actual); Status verified 2022-01

CONDITIONS: Aging Problems; Wrinkle
Keywords: Acupuncture; Thread embedding acupuncture; Aesthetic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Manual acupuncture (Active Comparator): The subjects/population of this study is woman at age 30-50 who meet the inclusion criteria. Subjects group with manual acupuncture treatment will be treated with 6 session of manual acupuncture at:
  From the superior of zygomatic arch through ST 2 to LI 20 bilaterally using a needle size of 0.25 x 60 mm From the inferior of zygomatic arch through SI 18 to ST 4 bilaterally using a needle size of 0.25 x 60 mm From ST 7 to ST 4 bilaterally using a needle size of 0.25 x 60 mm Along the nasolabial crease through ST 4 to the bilateral EXHN-8 using a needle size of 0.25 x 40 mm
  Interventions: Other: Manual acupuncture
- Thread embedding acupuncture (Active Comparator): The subjects/population of this study is woman at age 30-50 who meet the inclusion criteria. Subjects group with thread embedding acupuncture group treatment will be treated with 1 session of thread embedding acupuncture at:
  From the superior of zygomatic arch through ST 2 to LI 20 bilaterally using a gauge and length of the needle of 31G x 50 mm From the inferior of zygomatic arch through SI 18 to ST 4 bilaterally using a gauge and length of the needle of 31G x 50 mm From ST 7 to ST 4 bilaterally using a gauge and length of the needle of 31G x 50 mm Along the nasolabial crease through ST 4 to the bilateral EXHN-8 using a gauge and length of the needle of 31G x 30 mm
  Interventions: Other: Thread embedding acupuncture

INTERVENTIONS:
Other: Manual acupuncture — Manual acupuncture using filiform needle
  Arms: Manual acupuncture
Other: Thread embedding acupuncture — Thread Embedding acupuncture using Polydioxanone thread
  Arms: Thread embedding acupuncture

SUMMARY:
This study was aimed to compare the effectiveness of polydioxanone thread embedding acupuncture and manual acupuncture on the reduction of the nasolabial fold. One cycle of therapy in the manual acupuncture group (MA) was carried out with 6 sessions of manual acupuncture therapy while one cycle of therapy in the thread embedding acupuncture group (TEA) received 1 single session of thread embedding acupuncture. The outcome of the study was assessed based on the length of the nasolabial fold as measured by a digital vernier caliper, changes in wrinkle severity rating scale, and patient's subjective opinion of her nasolabial fold using visual analog scale. Outcome measurements were carried out after completing 1 cycle, and follow up at 2 weeks, 1 month, 2 months and 3 months after completing 1 cycle.

ELIGIBILITY:
Inclusion Criteria:

* Woman
* Age 30-50 years old
* WSRS scale 3 to 4
* Willing to follow the research to completion
* Subjects who do not have a history of filler injection and/implants, laser therapy, microdermabrasion, peeling, botulinum toxin therapy, manual acupuncture on the face, thread embedding acupuncture on the face and does not either oral or topically use collagen within 6 months
* Body mass index of ≥ 18.5
* Signed the informed consent

Exclusion Criteria:

* Subjects with facial muscle paralysis disorders
* Subjects with history of keloids and/or hypertrophic scars, subjects with tumors or infection or inflammation at the treatment area
* Subjects with allergies to stainless steel, PDO threads, topical anesthetics lidocaine
* Pregnant and lactating subjects
* Subjects with cancer
* Subjects with history of bleeding disorders or are taking anticoagulant or antiplatelet.
* Subjects suffering from fever (≥ 37.5°C), cough, fatigue
* Subjects with blood glucose POCT (Point of Care Testing) levels of ≥ 200 mg/dl

Ages: 30 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2021-09-08 (Actual); Primary Completion 2022-01-26 (Actual); Study Completion 2022-01-26 (Actual)

PRIMARY OUTCOMES:
Nasolabial fold length | Before intervention (baseline), after completing 1 cycle, at 2 weeks, 1 month, 2 month, and 3 month follow up
  Mean difference of nasolabial fold length (measured using digital vernier calipers in millimeters) between two groups
Wrinkle severity rating scale (WSRS) | Before intervention (baseline), after completing 1 cycle, at 2 weeks, 1 month, 2 month, and 3 month follow up
  Mean difference of WSRS between two groups

SECONDARY OUTCOMES:
Visual analog scale (VAS) | Before intervention (baseline), after completing 1 cycle, at 2 weeks, 1 month, 2 months, and 3 months follow up
  Mean difference of VAS (patient's subjective opinion of her nasolabial fold) between two groups

CONTACTS AND LOCATIONS:
Overall Officials: Yolanda Teja, Principal Investigator — Faculty of Medicine, University of Indonesia
Locations (1):
- Cipto Mangunkusumo Hospital, Jakarta Pusat, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: No